CLINICAL TRIAL: NCT03963089
Title: Effect of Tidal Volume Change on Pressure-based Prediction of Fluid Responsiveness in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1902-119-1013
Record Dates: First submitted 2019-05-19; First posted 2019-05-24 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Plasma Volume; Tidal Volume
Keywords: Fluid Therapy; Hemodynamic Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Measure pulse pressure variation and systolic pressure variation after each set of tidal volume to 6mL/kg, 10mL/kg and 14mL/kg. Measure respiratory variation of aortic blood flow peak velocity via transesophageal echocardiography at tidal volume of 10mL/kg.
  Measure stroke volume index via transesophageal echocardiography before and 5 min after fluid loading with 10mL/kg of crystalloid.
  Interventions: Procedure: Tidal volume_6mL/kg; Procedure: Tidal volume_10mL/kg; Procedure: Tidal volume_14mL/kg; Procedure: Fluid loading

INTERVENTIONS:
Procedure: Tidal volume_6mL/kg — Set tidal volume to 6mL/kg for 1 minute
Procedure: Tidal volume_10mL/kg — Set tidal volume to 10mL/kg for 1 minute
Procedure: Tidal volume_14mL/kg — Set tidal volume to 10mL/kg for 1 minute
Procedure: Fluid loading — Administer 10mL/kg of crystalloid for 5 minutes

SUMMARY:
This study evaluates predictability of fluid responsiveness of pressure-based dynamic variables such as pulse pressure variation and systolic pressure variation, according to tidal volume change in patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
Pressure-based dynamic variables such as pulse pressure variation(PPV) and systolic pressure variation(SPV) are known to be unreliable for prediction of fluid responsiveness in children.

The hypothesis is that tidal volume change in mechanically ventilated children undergoing anesthesia would affect reliability of aforementioned dynamic variables in prediction of fluid responsiveness, especially in the way that reliability increases for high tidal volume.

In children undergoing cardiac surgery, tidal volume is changed to 6mL/kg, 10mL/kg and 14mL/kg after closure of sternum, followed by measurement of PPV, SPV. We also measure the respiratory variation of aortic blood peak velocity(△Vpeak) via transesophageal echocardiography, which is known to best predict fluid responsiveness.

Afterward, 10mL/kg of crystalloid solution is administered for fluid loading. 'Fluid responder' is defined as subjects with increase of stroke volume index more than 15% after fluid loading of 10mL/kg.

With these data, whether the predictability of fluid responsiveness of PPV and SPV changes according to change in tidal volume is evaluated by comparing the area under the curve of the receiver-operating characteristics curve between themselves and △Vpeak.

ELIGIBILITY:
Inclusion Criteria:

* Children younger than 6 years old planned to undergo ventricular septal defect closure or atrial septal defect closure under general anesthesia

Exclusion Criteria:

* Children with other complex cardiac defects
* Children with arrhythmia
* Children with preoperatively measured ejection fraction of less than 30%
* Children with underlying pulmonary disease

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
Stroke volume index | From sternal closure to 5 minutes after fluid loading
  Define subject that shows increase of stroke volume index more than 15% after 10mL/kg of fluid loading as fluid responder, otherwise as non-responder
Predictability_PPV and SPV | From sternal closure to 5 minutes after fluid loading
  Area under the curve of the receiver-operative characteristic curve for prediction of fluid responder of pulse pressure variation and systolic pressure variation after each change of set tidal volume

SECONDARY OUTCOMES:
Predictability_△Vpeak | From sternal closure to 5 minutes after fluid loading
  Area under the curve of the receiver-operative characteristic curve for prediction of fluid responder of respiratory variation of aortic blood flow peak velocity measured via transesophageal echocardiography at tidal volume of 10mL/kg
Grey zone | From sternal closure to 5 minutes after fluid loading
  Compare the range that the prediction of fluid responsiveness is unreliable (grey zone) for each variable in each set tidal volume

OTHER OUTCOMES:
Heart rate | From start of anesthesia to end of anesthesia
  Heart rate determined by electrocardiogram (beats/min)
Pulse oximetry | From start of anesthesia to end of anesthesia
  Pulse oximetry determined by photoplethysmography (%)
End-tidal carbon dioxide | From start of anesthesia to end of anesthesia
  End-tidal carbon dioxide measured from ventilatory circuit (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, M.D, Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gan H, Cannesson M, Chandler JR, Ansermino JM. Predicting fluid responsiveness in children: a systematic review. Anesth Analg. 2013 Dec;117(6):1380-92. doi: 10.1213/ANE.0b013e3182a9557e. PMID 24257389
- [Background] Durand P, Chevret L, Essouri S, Haas V, Devictor D. Respiratory variations in aortic blood flow predict fluid responsiveness in ventilated children. Intensive Care Med. 2008 May;34(5):888-94. doi: 10.1007/s00134-008-1021-z. Epub 2008 Feb 8. PMID 18259726
- [Background] Byon HJ, Lim CW, Lee JH, Park YH, Kim HS, Kim CS, Kim JT. Prediction of fluid responsiveness in mechanically ventilated children undergoing neurosurgery. Br J Anaesth. 2013 Apr;110(4):586-91. doi: 10.1093/bja/aes467. Epub 2012 Dec 18. PMID 23250892
- [Background] Cannesson M, Le Manach Y, Hofer CK, Goarin JP, Lehot JJ, Vallet B, Tavernier B. Assessing the diagnostic accuracy of pulse pressure variations for the prediction of fluid responsiveness: a "gray zone" approach. Anesthesiology. 2011 Aug;115(2):231-41. doi: 10.1097/ALN.0b013e318225b80a. PMID 21705869
- [Background] Min JJ, Gil NS, Lee JH, Ryu DK, Kim CS, Lee SM. Predictor of fluid responsiveness in the 'grey zone': augmented pulse pressure variation through a temporary increase in tidal volume. Br J Anaesth. 2017 Jul 1;119(1):50-56. doi: 10.1093/bja/aex074. PMID 28974059